CLINICAL TRIAL: NCT06120140
Title: A Phase 2, Open-Label, Randomized Trial Evaluating the Impact of Enhanced Versus Standard Dermatologic Management on Selected Dermatologic Adverse Events Among Patients With Locally Advanced or Metastatic EGFR-Mutated NSCLC Treated First-Line With Amivantamab + Lazertinib
Brief Title: Enhanced Dermatological Care to Reduce Rash and Paronychia in Epidermal Growth Factor Receptor (EGRF)-Mutated Non-Small Cell Lung Cancer (NSCLC) Treated First-line With Amivantamab Plus Lazertinib
Acronym: COCOON
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61186372NSC2007; 61186372NSC2007 (Other: Janssen Research & Development, LLC); 2023-505863-35-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — amivantamab; lazertinib; Doxycycline; Minocycline; Clindamycin; Chlorhexidine; ruxolitinib; Tacrolimus; gluconic acid; Propranolol; Timolol; Clobetasol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A: Enhanced Dermatologic Management (Experimental): Participants will receive enhanced dermatologic management to reduce toxicities in skin and nail with doxycycline tablet or minocycline capsule, clindamycin topical lotion, chlorhexidine topical solution, and noncomedogenic skin moisturizer during background anticancer treatment of advanced or metastatic epidermal growth factor receptor (EGFR)-mutated non-small cell lung cancer (NSCLC) with amivantamab intravenously (Dose 1 for body weight [BW] less than 80 kilograms [kg] and Dose 2 for BW greater than or equal to [>=] 80 kg as IV infusion [Arm A]) until documented disease progression using Response Evaluation Criteria in Solid Tumors version 1.1).
  Interventions: Drug: Amivantamab IV; Drug: Lazertinib; Drug: Doxycycline; Drug: Minocycline; Drug: Clindamycin; Drug: Chlorhexidine; Other: Noncomedogenic skin moisturizer
- Arm B: Standard-of-Care Dermatologic Management (Active Comparator): Participants will receive standard care for dermatologic management according to local practice to reduce dermatologic toxicities in skin and nail during background anticancer treatment of advanced or metastatic EGFR-mutated NSCLC with amivantamab administered as IV infusion plus lazertinib, dose and dosing schedule as same as experimental arm.
  Interventions: Drug: Amivantamab IV; Drug: Lazertinib; Drug: Chlorhexidine; Other: Noncomedogenic skin moisturizer
- Sub-study: Cohort A: Ruxolitinib (Experimental): Participants enrolled in Arms A and B of the main study who experience new-onset or persistent specific DAEIs (Grade greater than or equal to [>=] 2, as defined by National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE] v5.0) will be enrolled and receive reactive treatment with ruxolitinib in the sub-study. Participants in the sub-study will continue to receive amivantamab and lazertinib.
  Interventions: Drug: Amivantamab IV; Drug: Lazertinib; Drug: Doxycycline; Drug: Minocycline; Drug: Clindamycin; Drug: Chlorhexidine; Other: Noncomedogenic skin moisturizer; Other: Ruxolitinib
- Sub-study: Cohort B: Tacrolimus (Experimental): Participants enrolled in Arms A and B of the main study who experience new-onset or persistent specific DAEIs (Grade >= 2, as defined by NCI-CTCAE v5.0) will be enrolled and receive reactive treatment with tacrolimus in the sub-study. Participants in the sub-study will continue to receive amivantamab and lazertinib.
  Interventions: Drug: Amivantamab IV; Drug: Lazertinib; Drug: Doxycycline; Drug: Minocycline; Drug: Clindamycin; Drug: Chlorhexidine; Other: Noncomedogenic skin moisturizer; Other: Tacrolimus
- Amivantamab Subcutaneous (SC) Expansion Cohort: Standard Schedule (Experimental): Participants will receive modified enhanced dermatologic management with oral doxycycline or minocycline, zinc gluconate and noncomedogenic skin moisturizer during background anticancer treatment of advanced or metastatic EGFR mutated NSCLC with amivantamab SC and lazertinib as per standard schedule. If a participant develops a dermatologic adverse event of interest (DAEI) they will receive early intervention as follows: for facial (ruxolitinib), for scalp (oral propranolol and clobetasol), for paronychia (chlorhexidine in addition to timolol) until documented disease progression using Response Evaluation Criteria in Solid Tumors version 1.1.
  Interventions: Drug: Amivantamab SC; Drug: Lazertinib; Drug: Doxycycline; Drug: Minocycline; Drug: Chlorhexidine; Other: Noncomedogenic skin moisturizer; Other: Ruxolitinib; Drug: Zinc gluconate; Drug: Propranolol; Drug: Timolol; Drug: Clobetasol
- Amivantamab SC Expansion Cohort: Modified Schedule (Experimental): Participants will receive modified enhanced dermatologic management with oral doxycycline or minocycline, zinc gluconate and noncomedogenic skin moisturizer during background anticancer treatment of advanced or metastatic EGFR mutated NSCLC with amivantamab SC and lazertinib as per modified schedule. If a participant develops a DAEI they will receive early intervention as follows: for facial (ruxolitinib), for scalp (oral propranolol and clobetasol), for paronychia (chlorhexidine in addition to timolol) until documented disease progression using Response Evaluation Criteria in Solid Tumors version 1.1.
  Interventions: Drug: Amivantamab SC; Drug: Lazertinib; Drug: Doxycycline; Drug: Minocycline

INTERVENTIONS:
Drug: Amivantamab IV — Amivantamab will be administered.
  Other Names: JNJ-61186372
  Arms: Arm A: Enhanced Dermatologic Management; Arm B: Standard-of-Care Dermatologic Management; Sub-study: Cohort A: Ruxolitinib; Sub-study: Cohort B: Tacrolimus
Drug: Amivantamab SC — Amivantamab will be administered as SC injection.
  Other Names: JNJ-61186372
  Arms: Amivantamab SC Expansion Cohort: Modified Schedule; Amivantamab Subcutaneous (SC) Expansion Cohort: Standard Schedule
Drug: Lazertinib — Lazertinib tablet will be administered orally.
  Other Names: JNJ-73841937
Drug: Doxycycline — Doxycycline tablet will be administered orally.
  Arms: Amivantamab SC Expansion Cohort: Modified Schedule; Amivantamab Subcutaneous (SC) Expansion Cohort: Standard Schedule; Arm A: Enhanced Dermatologic Management; Sub-study: Cohort A: Ruxolitinib; Sub-study: Cohort B: Tacrolimus
Drug: Minocycline — Minocycline capsule will be administered orally.
  Arms: Amivantamab SC Expansion Cohort: Modified Schedule; Amivantamab Subcutaneous (SC) Expansion Cohort: Standard Schedule; Arm A: Enhanced Dermatologic Management; Sub-study: Cohort A: Ruxolitinib; Sub-study: Cohort B: Tacrolimus
Drug: Clindamycin — Clindamycin lotion will be used as topical application on the scalp.
  Arms: Arm A: Enhanced Dermatologic Management; Sub-study: Cohort A: Ruxolitinib; Sub-study: Cohort B: Tacrolimus
Drug: Chlorhexidine — Chlorhexidine solution will be used as topical application on hands and feet.
  Arms: Amivantamab Subcutaneous (SC) Expansion Cohort: Standard Schedule; Arm A: Enhanced Dermatologic Management; Arm B: Standard-of-Care Dermatologic Management; Sub-study: Cohort A: Ruxolitinib; Sub-study: Cohort B: Tacrolimus
Other: Noncomedogenic skin moisturizer — Noncomedogenic skin moisturizer will be used as topical application.
  Arms: Amivantamab Subcutaneous (SC) Expansion Cohort: Standard Schedule; Arm A: Enhanced Dermatologic Management; Arm B: Standard-of-Care Dermatologic Management; Sub-study: Cohort A: Ruxolitinib; Sub-study: Cohort B: Tacrolimus
Other: Ruxolitinib — Ruxolitinib will be used to the affected skin area.
  Arms: Amivantamab Subcutaneous (SC) Expansion Cohort: Standard Schedule; Sub-study: Cohort A: Ruxolitinib
Other: Tacrolimus — Tacrolimus will be used as topical application to the affected skin area.
  Arms: Sub-study: Cohort B: Tacrolimus
Drug: Zinc gluconate — Zinc gluconate tablet will be administered.
  Arms: Amivantamab Subcutaneous (SC) Expansion Cohort: Standard Schedule
Drug: Propranolol — Propranolol tablet will be administered.
  Arms: Amivantamab Subcutaneous (SC) Expansion Cohort: Standard Schedule
Drug: Timolol — Timolol will be used to the affected skin area.
  Arms: Amivantamab Subcutaneous (SC) Expansion Cohort: Standard Schedule
Drug: Clobetasol — Clobetasol shampoo will be used on the scalp.
  Arms: Amivantamab Subcutaneous (SC) Expansion Cohort: Standard Schedule

SUMMARY:
The purpose of this study is to evaluate whether enhanced dermatologic management can reduce incidence of grade greater than or equal to (>=) 2 dermatologic adverse events of interest (DAEIs) when compared with standard-of-care skin management and with modified enhanced dermatologic management in participants with locally advanced or metastatic stage IIIB/C-IV epidermal growth factor receptor (EGFR)-mutated non-small cell lung cancer (NSCLC) treated first-line with amivantamab and lazertinib. The study also includes Expansion cohorts (in 2 different schedules) to evaluate enhanced dermatologic management and early intervention for DAEIs or paronychia, in participants receiving subcutaneous amivantamab and lazertinib. A substudy will enroll participants from Arms A and B who experience specific new-onset or persistent DAEIs (Grade >=2) during treatment with intravenous (IV) amivantamab and lazertinib. This substudy aims to assess the reactive use of dermatologic treatment strategies in these participants.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed, locally advanced or metastatic non-small cell lung cancer (NSCLC); Is treatment naive and not amenable to curative therapy including surgical resection or (chemo) radiation. Adjuvant or neoadjuvant therapy for Stage I, Stage II or Stage IIIA disease is allowed if last dose administered more than 12 months prior to the development of locally advanced or metastatic disease
* Have a tumor that harbors an epidermal growth factor receptor (EGFR) Exon 19del or Exon 21 L858R substitution, as detected by an Food and Drug Administration (FDA)-approved or other validated test in a clinical laboratory improvement amendments (CLIA)-certified laboratory (sites in the United States) or an accredited local laboratory (sites outside of the United States) in accordance with site standard-of-care
* A participant with asymptomatic or previously treated and stable brain metastases may participate in this study. Participants with a history of symptomatic brain metastases must have had all lesions treated as clinically indicated (that is, no current indication for further definitive local therapy). Any definitive local therapy to brain metastases must have been completed at least 14 days prior to randomization, and the participant can be receiving no greater than 10 milligram (mg) prednisone or equivalent daily for the treatment of intracranial disease
* Can have prior or concurrent second malignancy (other than the disease under study) which natural history or treatment is unlikely to interfere with any study endpoints, safety, or the efficacy of the study treatment(s). For the amivantamab SC expansion cohorts: Due to the increased risk of skin cancer with ruxolitinib, participants with any prior or concurrent skin malignancies will be excluded
* Sub-study: Participants must have new-onset or persistent (defined as non-responsive to standard of care [SoC]) Grade >=2 specific DAEIs of the scalp, face, or body, as defined by NCI-CTCAE Grading v5.0 for DAEIs (excluding paronychia)

Exclusion Criteria:

* History of uncontrolled illness, including but not limited to uncontrolled diabetes; ongoing or active infection (includes infection requiring treatment with antimicrobial therapy [participants will be required to complete antibiotics 1 week prior to starting background anticancer treatment] or diagnosed or suspected viral infection). For the amivantamab SC expansion cohorts, this includes active localized serious infections; active bleeding diathesis; impaired oxygenation requiring continuous oxygen supplementation; refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of background anticancer treatment or doxycycline/minocycline; psychiatric illness, social situation, or any other circumstances that would limit compliance with study requirements; any ophthalmologic condition that is clinically unstable; pre-existing skin condition that would prevent adequate evaluations of dermatologic toxicity, as determined by the investigator
* Medical history of interstitial lung disease (ILD), including drug-induced ILD or radiation pneumonitis
* Known allergy, hypersensitivity, or intolerance to the excipients of amivantamab, lazertinib, or to tetracyclines, doxycycline, minocycline, timolol*, ruxolitinib*, zinc*, corticosteroids* or their excipients or to any component of the enhanced dermatologic management (*for the amivantamab SC expansion cohorts)
* Participant has received any prior systemic treatment at any time for locally advanced stage III B/C or metastatic stage IV disease (adjuvant or neoadjuvant therapy for stage I, II or IIIA disease is allowed if last dose administered more than 12 months prior to the development of locally advanced or metastatic disease)
* Participant has an active or past medical history of leptomeningeal disease
* Sub-study: Participants who have received prior treatment for epidermal growth factor receptor (EGFR)-induced DAEIs with JAK inhibitors (for Cohort A) or calcineurin inhibitors (for Cohort B)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Grade Greater Than or Equal to (>=) 2 Dermatologic Adverse Events of Interest (DAEIs) Within 12 Weeks After Initiation of Anticancer Treatment | Up to 12 weeks after initiation of anticancer treatment
  Number of participants with Grade >= 2 DAEIs within 12 weeks after initiation of anticancer treatment based on National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE) Version (v) 5.0 will be reported. DAEIs includes rash, dermatitis acneiform, pruritus, skin fissures, acne, folliculitis, erythema, eczema, rash maculo-papular, skin exfoliation, skin lesion, skin irritation, dermatitis, rash erythematous, rash macular, rash popular, rash pruritic, rash pustular, dermatitis contact, dermatitis exfoliative generalized, drug eruption, dyshidrotic eczema, eczema asteatotic and paronychia. As per NCI CTCAE v 5.0, severity scale ranges from Grade 1 (mild) to Grade 5 (death). Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening, and Grade 5= death related to adverse event.

SECONDARY OUTCOMES:
Number of Participants With DAEIs by Severity Based on NCI-CTCAE v 5.0 | Up to 12 weeks after initiation of anticancer treatment
  Number of participants with DAEIs by severity based on NCI-CTCAE v 5.0 will be reported.
Number of Participants With Grade >=2 DAEIs Within 6 Months After Initiation of Anticancer Treatment Based on NCI-CTCAE v 5.0 | Up to 6 months after initiation of anticancer treatment
  Number of participants with Grade >=2 DAEIs within 6 months after initiation of anticancer treatment based on NCI-CTCAE v 5.0 will be reported.
Number of Grade >= 2 DAEI Per Participants | Up to 12 months
  Number of grade >= 2 DAEI per participants will be reported.
Time to First Occurrence of Grade >=2 DAEI | Up to 12 months
  Time to first occurrence of Grade >=2 DAEI will be reported.
Time to Resolution of Grade >= 2 DAEI | Up to 12 months
  Time to resolution of Grade >= 2 DAEI will be reported.
Number of Participants With Paronychia by Severity Based on NCI-CTCAE v 5.0 | Up to 6 months after initiation of anticancer treatment
  Number of participants with paronychia by severity based on NCI-CTCAE v 5.0 will be reported.
Number of Participants With Scalp Rash by Severity Based on NCI-CTCAE v 5.0 | Up to 12 months after initiation of anticancer treatment
  Number of participants with scalp rash by severity based on NCI-CTCAE v 5.0 will be reported.
Change From Baseline in Skindex Symptoms Domain Score up to 12 Months | Baseline, up to Month 12
  Change from baseline in skindex symptoms domain score up to 12 months will be reported. The score of quality of life will be assessed using the Skindex-16 questionnaire. Skindex-16 is used for participants to rate skin conditions.
Change From Baseline in Patient's Global Impression-Severity (PGI-S) Rash up to 12 Months | Baseline, up to Month 12
  Change from baseline in PGI-S rash up to 12 months will be reported. Participant quality of life will be evaluated using PGI-S Rash. PGI-S is a single-item questionnaire assessing participants disease severity on a 7-point response scale.
Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30) Score up to 12 Months | Baseline, up to Month 12
  Change from baseline in EORTC-QLQ-C30 score up to 12 months will be reported. EORTC-QLQ-C30 is a core 30-item questionnaire for evaluating the health-related quality of life (HRQoL) of participants participating in cancer clinical studies.
Change From Baseline in EuroQol 5 - Dimension (EQ-5D) Patient-reported Outcome (PRO) up to 12 Months (for Amivantamab Subcutaneous Expansion Cohort Only) | Baseline, up to Month 12
  The EQ-5D questionnaire is a brief, generic HRQOL assessment that can that can also be used to incorporate participant preferences into health economic evaluations. The EQ-5D questionnaire assesses HRQOL in terms of degree of limitation on 5 health dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and as overall health using a visual analog scale with response options ranging from 0 (worst imaginable health) to 100 (best imaginable health). Lower scores indicate worsening. EQ-5D scores include EQ-5D valuation index score (a weighted scoring of the 5 dimension scores with a possible range from 0 to 1), EQ-5D visual analog scale (VAS) is a vertical VAS with scores ranging from 0 (worst imaginable health) to 100 (perfect health), and EQ5D descriptive system scores (five scores reflecting each of the 5 EQ-5D health dimensions ranging from 0 [no limitation] to 4 [incapacity]).
Percentage of Participants With Dose Reductions, Dose Interruptions, and Dose Discontinuations of Anticancer Treatment due to DAEIs | Up to 12 months
  Percentage of participants with dose reductions, dose interruptions, and dose discontinuations of anticancer treatment due to DAEIs will be reported.
Relative Dose Intensity (RDI) of Anticancer Treatment | Up to 12 months
  Relative dose intensity of anticancer treatment will be reported. The relative dose intensity is defined as the ratio of total actually received dose versus total prescribed dose.
Percentage of Participants With Venous Thromboembolism (VTE) Adverse Events (AEs) by Severity Based on NCI-CTCAE v 5.0 | Up to 12 months
  Percentage of participants with VTE AEs (pulmonary embolism and deep vein thrombosis) by severity based on NCI-CTCAE v 5.0 will be reported. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.
Percentage of Participants With Adverse Events (AEs) by Severity Based on NCI-CTCAE v 5.0 | Up to 12 months
  Percentage of participants with AEs by severity based on NCI-CTCAE v 5.0 will be reported. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.
Progression Free Survival (PFS) | Up to 12 months
  PFS is defined as the time from the date of randomization to the date of first documented disease progression, as defined in the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, or death due to any cause, whichever occurs first.
Overall Response Rate (ORR) | Up to 12 months
  ORR is defined as the percentage of participants who achieve a partial response (PR) or better response using RECIST v1.1 as assessed by the investigator.
Duration of Response (DoR) | Up to 12 months
  DOR will be calculated among responders (with a PR or better response) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the RECIST v1.1 response criteria.
Amivantamab SC Expansion Cohorts: Number of Participants With Grade >= 2 DAEIs Within 12 Weeks After Initiation of Anticancer Treatment | Up to 12 weeks after initiation of anticancer treatment
  Participants with Grade >= 2 DAEIs within 12 weeks after initiation of anticancer treatment based on NCI-CTCAE v 5.0 will be reported. DAEIs includes rash, dermatitis acneiform, pruritus, skin fissures, acne, folliculitis, erythema, eczema, rash maculo-papular, skin exfoliation, skin lesion, skin irritation, dermatitis, rash erythematous, rash macular, rash popular, rash pruritic, rash pustular, dermatitis contact, dermatitis exfoliative generalized, drug eruption, dyshidrotic eczema, eczema asteatotic and paronychia. As per NCI-CTCAE v 5.0, severity scale ranges from Grade 1 (mild) to Grade 5 (death). Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening, and Grade 5= death related to adverse event.
Amivantamab SC Expansion Cohorts: Percentage of Participants With an Improvement in DAEI After Starting Early Intervention | Up to 12 months
  Percentage of participants showing an improvement in DAEI by a minimum of 1 NCI-CTCAE grade after starting early intervention will be reported. As per NCI-CTCAE v 5.0, severity scale ranges from Grade 1 (mild) to Grade 5 (death). Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening, and Grade 5= death related to adverse event.
Amivantamab SC Expansion Cohorts: Time to Improvement of DAEIs After Starting Early Intervention | Up to 12 months
  Time to improvement of DAEIs by a minimum of 1 NCI-CTCAE grade after starting early intervention will be reported. As per NCI-CTCAE v 5.0, severity scale ranges from Grade 1 (mild) to Grade 5 (death). Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening, and Grade 5= death related to adverse event.

OTHER OUTCOMES:
Percentage of Participants Achieving Best Response for the Dermatologic Adverse Event | Up to 12 weeks
  Participants achieving best response within 12 weeks of treatment defined as NCI-CTCAE level of the dermatologic adverse event improvement by at least 1 level will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (93):
- United States (28):
  - Ironwood Cancer and Research Center, Chandler, Arizona
  - City of Hope, Duarte, California
  - Providence Fullerton, Fullerton, California
  - Los Angeles Cancer Network, Glendale, California
  - City of Hope Seacliff, Huntington Beach, California
  - City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California
  - City of Hope Long Beach Elm, Long Beach, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - Keck Hospital of USC, Los Angeles, California
  - USC Norris Oncology Hematology Newport Beach, Newport Beach, California
  - Kaiser Permanente Oakland Medical Center, Oakland, California
  - Kaiser Permanente Roseville Medical Center, Roseville, California
  - Kaiser Permanente San Francisco Medical Center, San Francisco, California
  - Kaiser Permanente Santa Clara Medical Center, Santa Clara, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente Northern California, Vallejo, California
  - Kaiser Permanente Walnut Creek Medical Center, Walnut Creek, California
  - University Cancer & Blood Center, Athens, Georgia
  - Hope and Healing Care, Hinsdale, Illinois
  - Oncology Hematology Associates, Springfield, Missouri
  - Renown Health Medical Oncology, Reno, Nevada
  - Hunterdon Hematology Oncology, Flemington, New Jersey
  - Clinical Research Alliance Inc, Westbury, New York
  - Regional Medical Oncology Center, Wilson, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Valley Medical Center, Renton, Washington
  - Gundersen Health System, West Salem, Wisconsin
- Argentina (5):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - IADT Instituto Argentino de Diagnostico y Tratamiento, CABA
  - Centro Medico Austral, Capital Federal
  - Hospital Italiano de La Plata, La Plata
  - Hospital Privado de la Comunidad, Mar del Plata
- Brazil (11):
  - CTO Centro De Tratamento Oncologico LTDA, Belém
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Liga Paranaense de Combate ao Cancer, Curitiba
  - Fundacao Doutor Amaral Carvalho, Jaú
  - Hospital Nossa Senhora da Conceicao S A, Porto Alegre
  - Nucleo de Oncologia da Bahia Oncoclinicas, Salvador
  - Hospital Ana Nery Santa Cruz do Sul, Santa Cruz do Sul
  - Fundacao Faculdade de Medicina - Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
  - Servicos de Tratamento ao Cancer de Taubate LTDA - Instituto do Cancer Brasil Unidade Taubate, Taubaté
  - Associacao Feminina de Educacao e Combate ao Cancer Hospital Santa Rita de Cassia, Vitória
- China (11):
  - Changzhou No 2 Peoples Hospital, Changzhou
  - West China Hospital, Chengdoucun
  - Sichuan Cancer Hospital, Chengdu
  - The First Affiliated Hospital Sun Yat sen University, Guangzhou
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Harbin medical university cancer hospital, Harbin
  - Huizhou Municipal Central Hospital, Huizhou
  - Zhongda Hospital Southeast University, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
  - Henan Cancer Hospital, Zhengzhou
- France (3):
  - Hopital Nord, Marseille
  - Hopital PASTEUR, Nice
  - Institut Curie, Paris
- Germany (6):
  - Universitaetsklinikum der RWTH Aachen, Aachen
  - Kliniken Essen-Mitte, Essen
  - Universitaetsklinikum Giessen und Marburg GmbH, Giessen
  - Thoraxklinik am Universitatsklinikum Heidelberg, Heidelberg
  - Klinikum Kassel GmbH, Kassel
  - Universitaetsklinikum Schleswig Holstein Campus Kiel, Kiel
- Malaysia (4):
  - Hospital Pulau Pinang, George Town
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Hospital Umum Sarawak, Kuching
- South Korea (3):
  - Chungbuk National University Hospital, Cheongju-si
  - Gachon University Gil Hospital, Incheon
  - Severance Hospital Yonsei University Health System, Seoul
- Spain (9):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. Gral. Univ. de Alicante, Alicante
  - Hosp. Univ. Quiron Dexeus, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. de Jaen, Jaén
  - Hosp. Univ. Lucus Augusti, Lugo
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp Regional Univ de Malaga, Málaga
  - Hosp. Ntra. Sra. de Valme, Seville
- Taiwan (5):
  - Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan
  - National Taiwan University Hospital Hsin Chu Branch, Taoyuan District
- Turkey (Türkiye) (8):
  - Adana City Hospital, Adana
  - Gulhane Training and Research Hospital, Ankara
  - Gazi University Hospital, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Bakirkoy Training and Research Hospital, Istanbul
  - I A U VM Medical Park Florya Hastanesi, Istanbul
  - Ege University Medical Faculty, Izmir
  - Ondokuz Mayis University, Samsun

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency